CLINICAL TRIAL: NCT03953339
Title: Neuropathy of the Suprascapular Nerve Before and After Reconstruction of the Cuff
Acronym: Neurospura
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Balgrist University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NeuroW514
Record Dates: First submitted 2017-06-29; First posted 2019-05-16 (Actual); Last update posted 2019-05-16 (Actual); Status verified 2019-05

CONDITIONS: Cuff Rotator Full Thickness Tear; Cuff Rotator Syndrome
MeSH Terms: interventions — Drainage

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- no release (Active Comparator): no release of the suprascapular nerve during arthroscopic repair of a rotator cuff tendon repair
  Interventions: Procedure: Release or no release of the suprascapular nerve
- release (Experimental): arthroscopic release of the suprascapular nerve according to the established, standard technique during arthroscopic repair of a rotator cuff tendon repair
  Interventions: Procedure: Release or no release of the suprascapular nerve

INTERVENTIONS:
Procedure: Release or no release of the suprascapular nerve

SUMMARY:
The suprascapular nerve innervates the musculi supra- and infraspinatus, which, as part of the rotator cuff, allow lifting and external rotation in the shoulder joint. Damage to this nerve can lead to pain and functional deficit. Causes of injury are compression by bony / ligamentous anomalies, fracture sequelae and traction damage. In the literature, a (often subclinical) traction damage is increasingly claimed by a muscle retraction after rupture of the supra- and / or infraspinatus tendon as a cause of pain and functional disturbances. The retraction of the ruptured tendon-muscular unit is said to lead to traction damage of the nerve, which can be demonstrated by pathological EMG derivations. By repositioning the tendon to its outbreak site, the nerve is occasionally overstretched, so that individual authors propagate a routine nerve decompression as prophylaxis. In individual cases, a previously pathologic EMG result could be improved after reconstitution of an rotator cuff rupture. However, prospective studies are not available.

It is not known how often a nerve damage is present before a rotator cuff operation and it is not known how often the tendon repair leads to nerve damage or recovery of damage. It is not known whether the surgical nerve decompression is associated with reduced postoperative pain and what a profit or what risks bring about a routine decompression of the nerve to the patient. To answer this question, this prospective randomized study is to be carried out.

DETAILED DESCRIPTION:
On the basis of preoperative electromyography (EMG) and electroneurography (ENG), the investigators would like to determine the frequency of suprascapular neuropathy in ruptures of supra- and / or infraspinatus tendons and the risk factors for their presence.

In a ruptured rotator cuff, the muscle is partly retracted so much that the innervating nerve (suprascapular nerve) is stretched and has pathological neurological findings. The Investigators now want to analyze how the arthroscopic reconstruction of the nasal suprascapular nerve affects the pre-operative neuropathy. Does the pre-existing nerve recover by decompression (liberation) from surrounding / entangling tissue or does decompression have no influence on measurable neurology? Other patients with rotator cuff ruptures have normal neurological findings preoperatively despite severe retraction of the muscular / tendon unit. In these cases, the investigators are interested in whether the mobilization and reconstruction of the torn muscle / tendon unit leads to a neurologically measurable elongation of the nerve. This nerve stretching is a possible explanation for protracted postoperative pain. With the postoperative electrophysiological measurements we can quantify this nerve change.

The comparison between preoperative and postoperative neurology findings allows confirmation or refutation of our hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Informed Consent
* MRI diagnosis of partial or full thickness rotator cuff tear

Exclusion Criteria:

* Previous surgery
* Fatty muscle infiltration Goutallier stages III and IV
* Diabetes mellitus
* pregnancy
* unwillingness or contraindications for Magnetic resonance imaging
* unwillingness or contraindications to electrophysiological assessment
* substance abuse

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2019-02-18 (Actual); Study Completion 2019-02-18 (Actual)

PRIMARY OUTCOMES:
electromyographic assessment of suprascapular nerve function | preoperatively, change from preoperatively to 3 months and change from 3 to 12 months
  sharp waves, complex repetitive discharges and fasciculations in supra- and infraspinatus muscles. Presence or absence
electromyographic assessment of suprascapular nerve function | preoperatively, change from preoperatively to 3 months and change from 3 to 12 months
  motor latency to supra- and infraspinatus muscles milliseconds
electromyographic assessment of suprascapular nerve function | preoperatively, change from preoperatively to 3 months and change from 3 to 12 months
  conduction velocity (m/sec)

SECONDARY OUTCOMES:
Maximal daily pain on visual analog scale | preoperatively and change from preoperatively to 3 months and change from 3 to 12 months
  Measurement of pain using a visual analog scale 100 points maximal imaginable pain; 0 no pain
Active range of motion | preoperatively and change from preoperatively to 3 months and change from 3 to 12 months
  Measurement of active elevation, abduction external and internal rotation in degrees measured with a handheld goniometer.
Strength | preoperatively and change from preoperatively to 3 months and change from 3 to 12 months
  Isometric measurement of strength of shoulder abduction in pounds (1 pound represents 1 point in the scoring system)using a validated dynamometer

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Balgrist, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided